CLINICAL TRIAL: NCT06986746
Title: Effects of Planned Awareness Program on Knowledge Regarding Prevention of Hypertensive Crisis in Hypertensive Patients.
Brief Title: Awareness Program on Knowledge Regarding Prevention of Hypertensive Crisis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Rec/ 02053 Kainat Gul
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
Keywords: Knowledge; Hypertension crisis; Planned awareness program
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypertension Crisis Awareness Program (Experimental): Education materials-consist of description about hypertension crisis, symptoms, causes and preventive measures (emphasizing on healthy lifestyle and physical activity) with pictorial presentation.
  Interventions: Other: Hypertension Crisis Awareness Program

INTERVENTIONS:
Other: Hypertension Crisis Awareness Program — Education materials-consist of description about hypertension crisis, symptoms, causes and preventive measures (emphasizing on healthy lifestyle and physical activity) with pictorial presentation.

SUMMARY:
To determine the effect of planned awareness program on knowledge regarding prevention of hypertensive crisis in hypertensive patients. Current literature is mainly on hypertension (HTN) control limited accessible studies on hypertension crises but these studies lack the detailed awareness program regarding prevention of hypertension crisis in diagnosed hypertension patients.

DETAILED DESCRIPTION:
Hypertension crisis(elevation of BP to 180/110mmHg or greater) is the very extreme form of poorly controlled hypertension that can develop in individuals with known pre-existing HTN and in patients who are not aware that they have hypertension.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed hypertensive patients

Exclusion Criteria:

* Language barrier
* Not willing to participate
* Unable to understand teaching program

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Hypertension Crisis Knowledge | 2 weeks
  Changes from baseline to 2 weeks, after the intervention awareness program, assessed through Questionnaire for hypertension crisis knowledge assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MS-CPPT PhD*, Principal Investigator — Riphah International University
Locations (1):
- Combined Military Hospitals, Tarbela, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No